CLINICAL TRIAL: NCT05092009
Title: Lung Cancer Organoids and Patient Derived Tumor Xenografts
Acronym: IPON-3
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Lung Organoids
Record Dates: First submitted 2021-09-15; First posted 2021-10-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Histocompatibility Testing; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tumour tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patiens: There is only one arm in this trial
  Interventions: Other: Tissue and blood

INTERVENTIONS:
Other: Tissue and blood — Tissue and blood will be derived from patient during a standard of care procedure

SUMMARY:
Extra tissue will be taken from patient during a procedure in standard of care. Also, through an existing line, 10ml of extra blood will be drawn. From this material the investigator will try to establish matched normal and primary human lung cancer organoids.

DETAILED DESCRIPTION:
Lung (tumor) material obtained from biopsies or surgical resection material that is not needed by the pathologist for diagnosis (i.e. to stage the patient or to perform molecular diagnosis) will be collected and used for the generation of matched normal and lung cancer organoids and/or PDX.

Biopsy material: Patients with (suspected) lung cancer will undergo a bronchoscopy or endobronchial ultrasound guided transbronchial needle aspiration (EBUS/EUS-TBNA) bronchoscopy for the collection of a lung / lymph node biopsy. Biopsies are collected according to standard of care procedures for i.e. the initial diagnosis and staging of lung cancer, and molecular profiling of recurrent tumors. During the standard of care biopsy procedure, an extra biopsy (lung and/or lymph node) will be collected and used for the generation of lung (cancer) organoids:

* Bronchoscopy: biopsy-derived lung (tumor) tissue from endobronchial tumors
* EBUS/EUS-TBNA bronchoscopy: cytology-derived lung (tumor) cells from mediastinal lymph nodes

A 10 ml blood sample will only be collected at the moment blood must be drawn according to standard of care procedures or when the patient has received an intravenous drip. The patient therefore does not require to undergo additional procedures.

Resection material: Patients who are selected to undergo surgical removal of a primary lung cancer will be included. The (tumor) material that will be used to make organoids and PDX will be derived from remaining healthy and tumor tissue that is not needed for the pathologist to make a diagnosis, to stage the patient or to perform a molecular diagnosis. The patient therefore does not require to undergo additional treatments or procedures. A 10 ml blood sample will be collected at the moment blood must be drawn pre-operatively according to standard of care procedures or from the intravenous drip the patient will receive before start surgery. The patient therefore does not require to undergo additional procedures.

Collection of clinical data: Clinical data will be collected from existing standard of care data:

* Histology
* Date diagnosis lung cancer
* TNM classification (eight edition)
* If performed, molecular analysis data such as Epidermal Growth Factor Receptor (EGFR) mutation, Anaplastic Lymphoma Kinase (ALK) translocation, Kirsten Rat Sarcoma (KRAS) viral oncogene homolog mutation etc. (Type of test, results)
* PD-L1 status if available. If available, type of test and PD-L1%
* Type, dose, and date of treatment the patient received before and/or after the collection tumor biopsy (chemotherapy, radiotherapy, tyrosine kinase inhibitors, immunotherapy). If applicable, also the date and dose of all cycles.

ELIGIBILITY:
Inclusion Criteria:

* All patients selected to undergo primary surgical resection of a primary lung cancer. All types of resection are eligible, e.g. wedge resection, segmental resection, lobectomy, pneumonectomy.
* All patients with (suspected) lung cancer that will undergo a bronchoscopy or endobronchial ultrasound guided transbronchial needle aspiration (EBUS/EUS-TBNA) bronchoscopy.

Exclusion Criteria:

There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Lung cancer organoids | 1 year
  Establishing matched normal and primary human lung cancer organoids from patient-derived (tumor) tissue material by establishing long term culturing and bio-banking conditions for matched normal and primary lung cancer organoids from patient-derived lung (tumor) material. From these, we will In the established organoids we will:
  • the rate of proliferation and cell death (turnover) will be calculated
Lung cancer organoids | 1 year
  Establishing matched normal and primary human lung cancer organoids from patient-derived (tumor) tissue material by establishing long term culturing and bio-banking conditions for matched normal and primary lung cancer organoids from patient-derived lung (tumor) material. From these, we will In the established organoids we will:
  • the size distribution of the organoids
Lung cancer organoids | 1 year
  Establishing matched normal and primary human lung cancer organoids from patient-derived (tumor) tissue material by establishing long term culturing and bio-banking conditions for matched normal and primary lung cancer organoids from patient-derived lung (tumor) material. From these, we will In the established organoids we will:
  • determine the frequency of primary, secondary and tertiary organoid formation

SECONDARY OUTCOMES:
Oncogenetic drivers | 1 year
  To define oncogenic drivers in lung cancer organoids
Tumor heterogeneity | 1 year
  To investigate the stability of (epi-) genetic and phenotypic tumor heterogeneity of cultured organoids compared to a primary/secondary biopsy
Molecular biology | 1 year
  To predict sensitivity and to get insight in the molecular biology of the response to immunotherapy, radiotherapy, cytotoxic and targeted agents
Treatment response | 1 year
  To compare treatment response in normal lung organoids and lung cancer organoids
Xenografts | 1 year
  To establish and characterize patient-derived tumor xenografts
Therapeutic approaches | 1 year
  To test novel therapeutic approaches in lung cancer organoids and clinically relevant PDX models, including radiotherapy combined with hypoxia activated prodrugs and immunotherapies
Developing biomarkers | 1 year
  To develop biomarker(s) of tumor response to be able to select patients who will benefit from novel treatment strategies.
Analysing blood | 1 year
  To analyze (ct)DNA in organoid-derived culture supernatants and corresponding patient-derived blood samples
Analysing blood | 1 year
  To analyze metabolites in organoid-derived culture supernatants and corresponding patient-derived blood samples
Analysing blood | 1 year
  To analyze RNA in organoid-derived culture supernatants and corresponding patient-derived blood samples
Analysing blood | 1 year
  To analyze proteins in organoid-derived culture supernatants and corresponding patient-derived blood samples
Analysing blood | 1 year
  To analyze microvesicles secreted by lung cancer cells in organoid-derived culture supernatants and corresponding patient-derived blood samples

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Zuyderland Medical Center, Heerlen
  - Maastricht Radiation Oncology (Maastro), Maastricht
  - MUMC+, Maastricht

IPD SHARING:
Plan to Share IPD: No